CLINICAL TRIAL: NCT06286761
Title: Routine Validation and Reproducibility Testing of Laboratory Assays and Research Techniques Used for Metabolism Research
Brief Title: Routine Validation and Reproducibility Testing of Laboratory Measures and Research Techniques Used for Metabolism Research (VAL)
Acronym: VAL
Status: Recruiting | Type: Observational
Sponsor: Bettina Mittendorfer (Other)
Responsible Party: Sponsor-Investigator, Bettina Mittendorfer, Senior Associate Dean for Research; Professor, Medicine & Nutrition; NextGen Director of Clinical and Translational Sciences Unit, University of Missouri-Columbia
Organization: University of Missouri-Columbia (Other)
Other Study IDs: 2100332
Record Dates: First submitted 2024-02-12; First posted 2024-02-29 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Single arm: For blood assay validation and/or reproducibility testing, blood samples will be taken after an overnight fast or after oral glucose or a mixed meal and analyzed. Measurements will be made by: using different assays to determine best conditions of measurement, or repeat testing on different days. Endothelial cells will be collected from a 20-gauge intravenous catheter. One to six 0.025" J-wires will be sequentially inserted into the catheter. These measurements will allow us to determine: the reproducibility and variability of assays used, best timing of blood and endothelial cell collection and best blood volumes and endothelial cell collection wire passes to reliably perform routine assays. For imaging validation, algorithm development, and/or reproducibility testing, participants may undergo DEXA, MRI, or MRS testing to develop or improve analysis algorithms, to evaluate variability of the measurements, or testing different equipment that measure the same variable.
  Interventions: Other: endothelial cell collection

INTERVENTIONS:
Other: endothelial cell collection — Participants may opt to have testing performed including blood sampling, intravenous catheter placement with endothelial cell collection, oral glucose tolerance test, consuming a test meal, having imaging performed such as MRI, DEXA, MRS to investigate use of different assays, different sample treatment approaches to determine optimal conditions that produce the most accurate and reproducible results, and/or repeat testing on different days or with different equipment that measures the same variable.
  Other Names: MRI; DEXA; MRS; blood testing; mixed meal; oral glucose tolerance testing

SUMMARY:
The purpose of this research study is to validate (check the accuracy of) laboratory assays, intravenous catheter insertion, and equipment or devices and their reproducibility, which is necessary to perform high quality research on chronic diseases (obesity, pre-diabetes and type-2 diabetes, dyslipidemia, non-alcoholic fatty liver disease, cardiovascular disease, etc.), nutrition, and metabolism (the process by which a substance is handled in your body) at the University of Missouri. As technology changes and we start to use new testing methods, it is necessary to compare results from old tests, equipment and devices and new tests, equipment, or devices and the reproducibility of these measurements to make sure we are getting accurate results. Reproducibility means performing the same test more than once to see if the same results can be achieved each time.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 and ≤75 years of age
* body mass index ≥18.5 and ≤45 kg/m2
* Weight stable (i.e., ≤3% change)
* ≤150 min of structured exercise/week for at least 2 months before entering the study
* Blood glucose: < 126 mg/dl fasted, < 200 mg/dl with 2 hour oral glucose tolerance testing
* Hemoglobin A1C (HbA1C) ≤6.5%
* Dyslipidemia triglycerides ≥125 mg/dL
* No chronic kidney disease
* Not vegan or vegetarian or on high protein diet (e.g. Atkins) or supplements that are not allowed
* No intolerance or allergies to study diet ingredients
* No excessive alcohol or tobacco consumption

Exclusion Criteria:

* <18 and >75 years of age
* body mass index <18.5 or >45 kg/m2
* history of or current significant organ system dysfunction (e.g., heart disease, stroke, diabetes, cancer in remission for <5 years, dementia, chronic kidney disease)
* allergies or intolerances to meal ingredients, vegans or vegetarians
* use of medications that could confound the study outcomes (e.g., anti-inflammatories, immune modulators, etc)
* take dietary supplements (e.g., certain pre- and pro-biotics, fiber, fish oil supplements)
* engaged in regular structured exercise >150 min per week
* alcohol use disorder as defined by the National Institute of Alcohol Abuse and Alcoholism or use of controlled substances
* pregnant women
* persons who use tobacco
* prisoners
* the inability to grant voluntary informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: convenience population of volunteers in mid-Missouri region
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-05-08 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Validation and reproducibility testing for blood assays | through study completion, an average of 10 weeks
  insulin, C-peptide, glucagon, substrates (free fatty acids, glucose, ketone bodies) and biomarkers of substrate metabolism (e.g., cytokines and adipokines)
Validation and reproducibility testing for endothelial cell collection | through study completion, an average of 10 weeks
  endothelial cell quantity collected
Validation and reproducibility testing for mixed meal ingestion | through study completion, an average of 10 weeks
  tolerability and palatability of meal type (protein concentration, carbohydrate concentration)
Validation and reproducibility testing for glucose tolerance testing | through study completion, an average of 10 weeks
  glucose levels
Validation and reproducibility testing for DEXA | through study completion, an average of 10 weeks
  body composition analysis
Validation and reproducibility testing for MRI | through study completion, an average of 10 weeks
  body composition analysis
Validation and reproducibility testing for MRS | through study completion, an average of 10 weeks
  body composition analysis

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Mittendorfer, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri School of Medicine, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No